CLINICAL TRIAL: NCT02994147
Title: A Proof-of-Concept Study of AC-201 Controlled-Release Tablet (CR Tablet) in Patients With Hemophilic Arthropathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: TWi Biotechnology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-201CR-HA-001
Record Dates: First submitted 2016-12-09; First posted 2016-12-15 (Estimated); Last update posted 2020-07-09 (Actual); Status verified 2020-07

CONDITIONS: Hemophilic Arthropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): 1. Subjects will initiate blinded study medication at a once daily (QD) regimen for 4 weeks, then titrate to twice daily (BID) for the remainder of the 24-week blinded treatment period.
  2. At Week 24, subjects will discontinue blinded study medication and start open-label treatment with AC-201CR. All subjects will initiate open-label AC-201CR QD for 4 weeks, then titrate to BID for the remainder of the study.
  Interventions: Drug: Placebo
- AC-201CR 72mg (Experimental): 1. Subjects will initiate blinded study medication at a once daily (QD) regimen for 4 weeks, then titrate to twice daily (BID) for the remainder of the 24-week blinded treatment period.
  2. At Week 24, subjects will discontinue blinded study medication and start open-label treatment with AC-201CR. All subjects will initiate open-label AC-201CR QD for 4 weeks, then titrate to BID for the remainder of the study.
  Interventions: Drug: AC-201CR

INTERVENTIONS:
Drug: Placebo — Placebo-only control study medication is the same formulation as active treatment without active ingredient
  Arms: Placebo
Drug: AC-201CR — The investigational product is formulated as controlled-release (CR) tablets
  Arms: AC-201CR 72mg

SUMMARY:
Repeated joint bleeding leads to hemophilic arthropathy (HA), which manifests with chronic synovitis, cartilage damage and bony destruction. Currently available treatments of HA, including analgesics, NSAIDs, and hyaluronic acid, are predominantly directed toward the symptomatic relief of pain and inflammation, with no or little effect on joint cartilage degeneration. AC201CR, a control released formulation of AC-201, demonstrates anti-inflammatory effects by reducing NLRP3 inflammasome assembly. AC-201 is also unique in that it influences both the anabolism and catabolism of chondrocytes in vitro and has shown cartilage-sparing properties in animal studies. The study is designed to evaluate the joint structure-modifying and symptom-relieving effects, safety, and tolerability of AC-201CR in subjects with HA.

ELIGIBILITY:
Inclusion Criteria:

1. Male age 20 to 65 years, inclusive
2. Diagnosis of Hemophilia A or B
3. Clinical diagnosis of hemophilic arthropathy in the knee(s) for at least 6 months
4. Pettersson score (based on X-ray) of 0 to 4 in at least one knee within 1 year of screening
5. IPSG (2012) overall score of 3 to 9 (based on MRI) in at least one knee at screening
6. Is able to read, understand, and sign the Informed Consent Form (ICF), communicate with the investigator, complete study diaries, and understand and comply with protocol requirements

Exclusion Criteria:

1. Total knee replacement in the primary knee
2. Presence of joint infections in the primary knee
3. Knee surgery within 6 months prior to screening in the primary knee
4. Intra-articular hyaluronic acid (IAHA) or platelet-rich plasma (PRP) injection in the primary knee within 6 months prior to screening
5. Use of any of the following medications after the screening visit:

   1. NSAID injection (oral NSAIDs including COX-2 inhibitors allowed)
   2. Glucosamine or chondroitin
6. History of high responder inhibitory antibodies to factor VIII or factor IX clotting factor, with titer >5 Bethesda units (BU), OR clinical evidence for presence of factor inhibitor
7. History of rheumatoid arthritis or gouty arthropathy
8. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) concentration >2x the upper limit of laboratory normal range (ULN), or bilirubin >1.5x ULN at screening
9. Positive test for human immunodeficiency virus (HIV), hepatitis B virus (HBV), or TB

Ages: 20 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-03-21 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-10-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline in IPSG (MRI) score for primary knee | 24 Weeks
  Knee arthropathy will be evaluated according to the 2012 IPSG (International Prophylaxis Study Group) rating scale. This scale is an additive scale with maximum value up to 17 points, comprising 2 subscores of soft tissue changes (maximum 9 points) and osteochondral changes (maximum 8 points).

SECONDARY OUTCOMES:
Change from baseline in IPSG (MRI) score for non-primary knee | 24 Weeks
Change from baseline in IPSG score by knee | 48 Weeks
Change from baseline in IPSG component scores by knee | 24 Weeks and 48 Weeks
Change from baseline in MRI-measured synovial thickness by knee | 24 Weeks and 48 Weeks
Change from baseline in ultrasonographic synovial thickness by knee | 24 Weeks and 48 Weeks
Change from baseline in ultrasonographic hyperemia score by knee | 24 Weeks and 48 Weeks
Change from baseline in knee pain (by VAS) by knee | 4, 12, 24, 28, 36 and 48 Weeks
Change from baseline in Short Form-36 score | 24 Weeks and 48 Weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No